CLINICAL TRIAL: NCT04112745
Title: The Effect of Magnetic Therapy on Pain Relief in Postoperation Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CMUH108-REC2-092
Record Dates: First submitted 2019-09-29; First posted 2019-10-02 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Surgical Patients; Hospitalized Patients
Keywords: Complementary Therapy; Static Magnet; Pain Relief; Hospitalized Patients

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental)
  Interventions: Other: Static magnet
- Control group (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Static magnet — Static magnet with 2,000 Gauss
  Arms: Experimental group
Other: Placebo — Polyvinyl chloride resin material black jewelry
  Arms: Control group

SUMMARY:
Using Complementary therapies with conventional treatments to relieve pain can reduce the patient's medical expenses and increase the patient's psychological feeling of self-control of the body. Static magnetic therapy is one of the non-invasive complementary therapies. The aim of this study was to explore the effect of static magnetic therapy on pain relief in hospitalized patients.

In this study, a quasi-experimental design with double-blind randomization method was proposed. 220 inpatients in a teaching hospital in central Taiwan were selected as the research subjects, and divided into experimental group and control group of 110. SPSS software package was used for descriptive and inferential statistical analysis in this study. For descriptive statistical analysis, frequency distribution, percentage, mean, and standard deviation were utilized. Inferential statistical analysis was applied with Chi-square test, Pearson's correlation, t-test, ANOVA, and Generalized Estimating Equations (GEE). The P value of significance level was set less than 0.05.

DETAILED DESCRIPTION:
Research Motivation and Research Issues:

The National Institutes of Health proposed six important strategies for pain management: studying the characteristics and needs of pain populations, prevention and care, identifying barriers and exclusions for pain care, providing individual pain care, professional education and training, and public awareness and communication. 80-100% of surgical patients experienced acute pain after surgery, and about 61-92% of postoperative patients experienced moderate or severe pain, and less than half of patients undergoing surgery showed that postoperative pain were alleviated. In the emergency treatment of musculoskeletal trauma patients, 40.9% of patients received medication. After pain treatment, only 12.5% of patients felt pain relief, and 23% of patients still felt moderate to severe pain when they left the emergency department. When pain is not properly relieved, it will have a negative impact on the patient, including quality of life and recovery of physical function, risk of complications, and even ineffective communication between doctors and patients. Proper pain assessment and care by caregivers can affect the effectiveness of pain relief in patients. Complementary therapy, in combination with conventional medicine, is one of the effective ways to relieve pain by reducing drug and medical costs and increasing the patient's self-care and autonomy. Complementary therapies can be divided into three broad categories: the first is natural products that are ingested through inhalation, external use or oral intake, including herbs, vitamins, minerals and probiotics. The second category is physical and mental interventional therapy, including art therapy, cognitive therapy, prayer, chanting, meditation, and energy complementary therapy, such as magnetic energy therapy. The third category is other categories such as local traditional therapy, Ayurvedic medicine, traditional Chinese medicine, homeopathy and natural remedies.

Magnetic therapy is a form of energy complementary therapy, which is the use of magnetic energy to produce energy for the relief or healing of diseases, usually divided into static magnetic therapy and dynamic electromagnetic therapy. In the implementation of magnetic therapy, there is no invasive treatment of pain and discomfort, no damage, so it is easy to be accepted by the public. The U.S. and Canada spend more than $500 million on static magnetic therapy to relieve pain, and global consumer spending exceeds $5 billion. The magnetic field has the effect of two distinct magnetic poles. The positive magnetic pole effect has the functions of oxidation, activation, excitation and pressure increase, and the negative magnetic pole effect has the functions of reduction, alkalization, relaxation, sedation and pressure resistance. Most of the research literature didn't show magnetic poles.

Therefore, this study focuses on the effect of magnetic complementary therapy on pain relief, in order to explore the magnetic therapy method and effect of pain relief.

Research design:

In this study, we adopted a double-blind randomized research design to investigate the effectiveness of magnetic complementary therapy in relieving pain in hospitalized patients. The outcomes of experimental group and the control group were repeatedly measured. Both groups received routine care and pain relief treatment, but the interventions were different: the participants of experimental group was adhered with magnets, and the control group with placebo.

Participants are randomly assigned to the experimental group and the control group, and the magnets or placebos are placed into the zipper bag and marked with serial numbers 1 to 100. When the cases are conducted in the study, the researchers take out the serial number zipper bag and paste it to the serial number. After the data collection, the researchers will identify the experimental and the control group according to the random table and the study case number.

The intervention materials are pre-packaged. Because the intervention materials (magnet and placebo) look exactly the same, none of the study subjects, the researchers who perform the sticking intervention material, and the physiological indicators monitoring were aware of the study case as an experimental group or a control group.

Interventions are implemented by the personnel including 1. Material assemblers: After a list of random numbers will be calculated by the randomizer, four pieces of magnets or placebos are arranged in each bag according to the random number table. 2. Magnet/placebo adhesion and evaluator: intervention adhesion and assessment of physiological indicators and rhythm variation measurements.

Research steps:

1. Screening for eligible cases.
2. Random assignment to the experimental group and the control group.
3. Pretest data collection: Pretest data collection is performed the day before surgery.
4. Day of surgery: According to the medical records, the researchers fill in the disease characteristics, including the name of the operation, the surgical site, the indwelling of the tube, and the total length of the wound. According to the case number, the magnet or the placebo, is pasted to the corresponding position of the healthy side limb.
5. On the first and second days after surgery, posttest data collection will be performed, including pain sensations: concise pain scale and anxiety scale; physiological indicators assessment and heart rhythm variation assessment.
6. On the 3rd day after surgery, the intervention material will be removed and posttest data will be collected. The researchers use the random table and the case number to identify the experimental and the control group.

Data analysis methods:

The collected quantitative data are encoded and analyzed by SPSS 24.0 statistical software package. According to the research variable attributes, the distributions of the independent variables and the dependent variables are verified by descriptive statistics, including the frequency distribution, percentage, average, and standard deviation. Inferential statistical analysis are applied with Chi-square test, Pearson's correlation, t-test, ANOVA, and Generalized Estimating Equations (GEE). The P value of significance level was set less than 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Prepare for surgery for adults.
2. The communicator is clear in Mandarin and Taiwanese.
3. Those who are willing to participate in this study and sign a consent form.
4. The patient has no history of arrhythmia or severe cardiopulmonary disease.
5. No allergies to adhesive fixtures.

Exclusion Criteria:

1. Patients with cancer or chronic pain that lasts for more than 6 months.
2. Those with effects on the accuracy of autonomic nervous system measurements: such as autonomic neuropathy.
3. Patients with excessive anxiety and nervousness who are unable to cooperate with the study.
4. A person who abuses painkillers or narcotic drugs.
5. Patients use electromagnetic medical supplies such as heart rhythms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain scale | Baseline, end of surgery, up until 3 days after surgery.
  The pain scale was calculated according to Brief Pain Inventory Short Form (BPI).
  The evaluation score was 0-10 points, with 0 being no pain and 10 being the worst pain. The classification scheme for average pain was 0-3 for mild, 4-6 for moderate, and 7-10 for severe.
Anxiety scale | Baseline, end of surgery, up until 3 days after surgery.
  The anxiety scale was calculated according to Hospital Anxiety and Depression Scale- Anxiety (HADS-A) which contained 7 items. This scale took the Likert scoring method, scoring 0-3, 0 points for never, 3-point for always. The score range was 0-21 points. A higher score indicated more anxious. The classification scheme for average anxiety was 0-7 for no anxiety, 8-10 for mild, 11-14 for moderate, and 15-21 for severe.

SECONDARY OUTCOMES:
heart rhythm variation | Baseline, end of surgery, up until 3 days after surgery.
  After lying flat for 10 minutes, take a 5-minute heart rate change measurement. Due to the measurement of time, mood and position will affect the variability of heart rhythm.

CONTACTS AND LOCATIONS:
Overall Officials: Shwn-Huey Shieh, PhD, Study Chair — China Medical University Hospital
Locations (1):
- China Medical University, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akin-Akinyosoye K, Frowd N, Marshall L, Stocks J, Fernandes GS, Valdes A, McWilliams DF, Zhang W, Doherty M, Ferguson E, Walsh DA. Traits associated with central pain augmentation in the Knee Pain In the Community (KPIC) cohort. Pain. 2018 Jun;159(6):1035-1044. doi: 10.1097/j.pain.0000000000001183. PMID 29438225
- [Background] Albuquerque WW, Costa RM, Fernandes Tde S, Porto AL. Evidences of the static magnetic field influence on cellular systems. Prog Biophys Mol Biol. 2016 May;121(1):16-28. doi: 10.1016/j.pbiomolbio.2016.03.003. Epub 2016 Mar 11. PMID 26975790
- [Background] Apfelbaum JL, Chen C, Mehta SS, Gan TJ. Postoperative pain experience: results from a national survey suggest postoperative pain continues to be undermanaged. Anesth Analg. 2003 Aug;97(2):534-540. doi: 10.1213/01.ANE.0000068822.10113.9E. PMID 12873949
- [Background] Barnes PM, Bloom B, Nahin RL. Complementary and alternative medicine use among adults and children: United States, 2007. Natl Health Stat Report. 2008 Dec 10;(12):1-23. PMID 19361005
- [Background] Brown CS, Ling FW, Wan JY, Pilla AA. Efficacy of static magnetic field therapy in chronic pelvic pain: a double-blind pilot study. Am J Obstet Gynecol. 2002 Dec;187(6):1581-7. doi: 10.1067/mob.2002.128026. PMID 12501067
- [Background] Cepeda MS, Carr DB, Sarquis T, Miranda N, Garcia RJ, Zarate C. Static magnetic therapy does not decrease pain or opioid requirements: a randomized double-blind trial. Anesth Analg. 2007 Feb;104(2):290-4. doi: 10.1213/01.ane.0000230613.25754.08. PMID 17242082
- [Background] Chou R, Gordon DB, de Leon-Casasola OA, Rosenberg JM, Bickler S, Brennan T, Carter T, Cassidy CL, Chittenden EH, Degenhardt E, Griffith S, Manworren R, McCarberg B, Montgomery R, Murphy J, Perkal MF, Suresh S, Sluka K, Strassels S, Thirlby R, Viscusi E, Walco GA, Warner L, Weisman SJ, Wu CL. Management of Postoperative Pain: A Clinical Practice Guideline From the American Pain Society, the American Society of Regional Anesthesia and Pain Medicine, and the American Society of Anesthesiologists' Committee on Regional Anesthesia, Executive Committee, and Administrative Council. J Pain. 2016 Feb;17(2):131-57. doi: 10.1016/j.jpain.2015.12.008. PMID 26827847
- [Background] Cowen SL, Phelps CE, Navratilova E, McKinzie DL, Okun A, Husain O, Gleason SD, Witkin JM, Porreca F. Chronic pain impairs cognitive flexibility and engages novel learning strategies in rats. Pain. 2018 Jul;159(7):1403-1412. doi: 10.1097/j.pain.0000000000001226. PMID 29578947
- [Background] de Heer EW, Ten Have M, van Marwijk HWJ, Dekker J, de Graaf R, Beekman ATF, van der Feltz-Cornelis CM. Pain as a risk factor for common mental disorders. Results from the Netherlands Mental Health Survey and Incidence Study-2: a longitudinal, population-based study. Pain. 2018 Apr;159(4):712-718. doi: 10.1097/j.pain.0000000000001133. PMID 29252911
- [Background] Eccles NK. A critical review of randomized controlled trials of static magnets for pain relief. J Altern Complement Med. 2005 Jun;11(3):495-509. doi: 10.1089/acm.2005.11.495. PMID 15992236
- [Background] Eghbali MEKR, Abazari P. Patients' viewpoints concerning post-surgical pain management. Iranian Journal of Nursing and Midwifery Research, 11(2), 2010
- [Background] Gan TJ, Habib AS, Miller TE, White W, Apfelbaum JL. Incidence, patient satisfaction, and perceptions of post-surgical pain: results from a US national survey. Curr Med Res Opin. 2014 Jan;30(1):149-60. doi: 10.1185/03007995.2013.860019. Epub 2013 Nov 15. PMID 24237004
- [Background] Haghighi MJ, Shahdadi H, Moghadam MP, Balouchi A. The Impact of Evidence-Based Practices on Postoperative Pain in Patients undergoing Gastrointestinal Surgery in Amiralmomenin Hospital in Zabol During 2014-2015. J Clin Diagn Res. 2016 Jul;10(7):IC01-IC04. doi: 10.7860/JCDR/2016/20961.8119. Epub 2016 Jul 1. PMID 27630865
- [Background] Hashimoto Y, Kawasumi M, Saito M. Effect of static magnetic field on cell migration. Electrical Engineering in Japan, 160(2), 46-52, 2007
- [Background] Hussain A, Erdek M. Interventional pain management for failed back surgery syndrome. Pain Pract. 2014 Jan;14(1):64-78. doi: 10.1111/papr.12035. Epub 2013 Feb 3. PMID 23374545
- [Background] Jaberi FM, Keshtgar S, Tavakkoli A, Pishva E, Geramizadeh B, Tanideh N, Jaberi MM. A moderate-intensity static magnetic field enhances repair of cartilage damage in rabbits. Arch Med Res. 2011 May;42(4):268-73. doi: 10.1016/j.arcmed.2011.06.004. PMID 21820604
- [Background] Kotani H, Kawaguchi H, Shimoaka T, Iwasaka M, Ueno S, Ozawa H, Nakamura K, Hoshi K. Strong static magnetic field stimulates bone formation to a definite orientation in vitro and in vivo. J Bone Miner Res. 2002 Oct;17(10):1814-21. doi: 10.1359/jbmr.2002.17.10.1814. PMID 12369785
- [Background] Lyle DB, Fuchs TA, Casamento JP, Davis CC, Swicord ML. Intracellular calcium signaling by Jurkat T-lymphocytes exposed to a 60 Hz magnetic field. Bioelectromagnetics. 1997;18(6):439-45. doi: 10.1002/(sici)1521-186x(1997)18:63.0.co;2-3. PMID 9261541
- [Background] Meulders A, Boddez Y, Blanco F, Van Den Houte M, Vlaeyen JWS. Reduced selective learning in patients with fibromyalgia vs healthy controls. Pain. 2018 Jul;159(7):1268-1276. doi: 10.1097/j.pain.0000000000001207. PMID 29533384
- [Background] Mogilner AY. Quality and cost-effectiveness of interventional pain procedures: minimally invasive lumbar decompression (MILD) as a paradigm? Pain Med. 2013 May;14(5):613-4. doi: 10.1111/pme.12140. Epub 2013 May 10. No abstract available. PMID 23663290
- [Background] Munn Z, Moola S, Riitano D, Lisy K. The development of a critical appraisal tool for use in systematic reviews addressing questions of prevalence. Int J Health Policy Manag. 2014 Aug 13;3(3):123-8. doi: 10.15171/ijhpm.2014.71. eCollection 2014 Aug. PMID 25197676
- [Background] Nettina SM, Msn A-B, Nettina SM. Lippincott manual of nursing practice: Lippincott Williams & Wilkins, 2013
- [Background] Pierik JG, IJzerman MJ, Gaakeer MI, Berben SA, van Eenennaam FL, van Vugt AB, Doggen CJ. Pain management in the emergency chain: the use and effectiveness of pain management in patients with acute musculoskeletal pain. Pain Med. 2015 May;16(5):970-84. doi: 10.1111/pme.12668. Epub 2014 Dec 28. PMID 25546003
- [Background] Ross SM. Combined DC and ELF magnetic fields can alter cell proliferation. Bioelectromagnetics. 1990;11(1):27-36. doi: 10.1002/bem.2250110105. PMID 2346505
- [Background] Sakurai T, Terashima S, Miyakoshi J. Enhanced secretion of prostaglandin E2 from osteoblasts by exposure to a strong static magnetic field. Bioelectromagnetics. 2008 May;29(4):277-83. doi: 10.1002/bem.20392. PMID 18163441
- [Background] Salomonowitz G, Friedrich M, Guntert BJ. [Medical relevance of magnetic fields in pain therapy]. Schmerz. 2011 Apr;25(2):157-60, 162-5. doi: 10.1007/s00482-010-1005-0. German. PMID 21258821
- [Background] Sieber FE, Barnett SR. Preventing postoperative complications in the elderly. Anesthesiol Clin. 2011 Mar;29(1):83-97. doi: 10.1016/j.anclin.2010.11.011. Epub 2011 Jan 5. PMID 21295754
- [Background] Simon LS. Relieving pain in America: A blueprint for transforming prevention, care, education, and research. Journal of pain & palliative care pharmacotherapy, 26(2), 197-198, 2012
- [Background] Stochkendahl MJ, Sorensen J, Vach W, Christensen HW, Hoilund-Carlsen PF, Hartvigsen J. Cost-effectiveness of chiropractic care versus self-management in patients with musculoskeletal chest pain. Open Heart. 2016 May 4;3(1):e000334. doi: 10.1136/openhrt-2015-000334. eCollection 2016. PMID 27175285
- [Background] Waxman SG, Cummins TR, Dib-Hajj SD, Black JA. Voltage-gated sodium channels and the molecular pathogenesis of pain: a review. J Rehabil Res Dev. 2000 Sep-Oct;37(5):517-28. PMID 11322150
- [Background] Weintraub MI, Wolfe GI, Barohn RA, Cole SP, Parry GJ, Hayat G, Cohen JA, Page JC, Bromberg MB, Schwartz SL; Magnetic Research Group. Static magnetic field therapy for symptomatic diabetic neuropathy: a randomized, double-blind, placebo-controlled trial. Arch Phys Med Rehabil. 2003 May;84(5):736-46. doi: 10.1016/s0003-9993(03)00106-0. PMID 12736891